CLINICAL TRIAL: NCT06320275
Title: Examining the Effect of Digital Storying on Fathers' Breastfeeding Self-efficiency
Brief Title: Fathers' Breastfeeding Self-efficiency
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cukurova University (Other)
Responsible Party: Principal Investigator, Elif DAĞLI, Principal Investigator, Cukurova University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: self-efficiency
Record Dates: First submitted 2023-12-15; First posted 2024-03-20 (Actual); Last update posted 2024-03-20 (Actual); Status verified 2024-03

CONDITIONS: FATHER; BREASTFEEDING
MeSH Terms: conditions — Breast Feeding | interventions — Control Groups

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Storytelling Intervention (Experimental): The Storytelling video intervention created is approximately 20 minutes long.
  Interventions: Behavioral: Storytelling Intervention
- control group (Active Comparator): Routine hospital protocol was applied to the women in this group. Storytelling fertility awareness video intervention was also given to the control group after the study.
  Interventions: Behavioral: Storytelling Intervention

INTERVENTIONS:
Behavioral: Storytelling Intervention — A storytelling fertility awareness video intervention, approximately 10 minutes in length, guided by a situation-specific theoretical framework and storytelling/narrative communication theory, was developed by the researchers.
  Other Names: control group

SUMMARY:
The purpose of this study was planned to examine the effect of the education given through digital storytelling method on fathers' breastfeeding self-efficacy perception. The research is in a quasi-experimental design with no pretest-posttest control group.

DETAILED DESCRIPTION:
In the study, intervention and control group data will be collected using the Personal Information Collection Form and the Father Breastfeeding Self-Efficacy Scale.

Personal Information Form: The Personal Information Form was developed by the researchers in line with literature information. There are questions about the socio-demographic characteristics of fathers, the role and responsibilities of fathers during breastfeeding.

Breastfeeding Self-Efficacy Scale for Fathers Short Form: The Breastfeeding Self-Efficacy Scale for Fathers was created by Dennis et al. to measure fathers' self-efficacy in supporting their spouses in breastfeeding, and its Cronbach's alpha value is 0.92.

ELIGIBILITY:
Inclusion Criteria:

* Not being between 0-6 weeks postpartum, not being married, not being literate

Exclusion Criteria:

-

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2023-02-01 (Actual); Primary Completion 2023-05-30 (Actual); Study Completion 2023-07-30 (Actual)

PRIMARY OUTCOMES:
Breastfeeding Self-Efficacy Scale for Fathers Short Form | up to 12 months
  Paternal Breastfeeding Self-Efficacy Scale- Short Form (Paternal BSES-SF): Paternal BSES-SF was developed by Dennis et al. (2018) to measure paternal self-efficacy in supporting their wives in breastfeeding and Cronbach's alpha value was 0.92. A Turkish validity-reliability study was conducted by Küçükoğlu (2022) and Cronbach's alpha value was found to be 0.93. The scale was applied to all fathers with newborn and breastfed infants and consisted of a single dimension with 14 items evaluated on a 5-point Likert scale (1=never 2=sometimes 3=sometimes 4=often 5=always). There are no reverse scored items in the scale. The minimum score to be obtained from the scale is 14 and the maximum score is 70. The cut-off point of the scale has not been determined,higher scores indicate higher confidence.

CONTACTS AND LOCATIONS:
Locations (3):
- Turkey (Türkiye) (3):
  - Cukurova University, Adana, Balcalı
  - Çukurova, Adana, Balcalı
  - Çukurova University, Adana

IPD SHARING:
Plan to Share IPD: No